CLINICAL TRIAL: NCT06298552
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase 3, Parallel-Group Design Study Evaluating the Efficacy and Safety of Efgartigimod IV in Adult Participants With Acetylcholine Receptor Binding Antibody Seronegative Generalized Myasthenia Gravis
Brief Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Efgartigimod IV in Patients With Acetylcholine Receptor Binding Antibody Seronegative Generalized Myasthenia Gravis
Acronym: ADAPT SERON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARGX-113-2308; 2024-511796-15-00 (Other: CTIS number)
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Generalized Myasthenia Gravis; gMG; Myasthenia Gravis, Generalized; Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV (Experimental): Patients receiving efgartigimod IV in both part A and part B
  Interventions: Biological: Efgartigimod IV
- Placebo (Placebo Comparator): Patients receiving placebo during part A and receiving efgartigimod IV during part B
  Interventions: Biological: Efgartigimod IV; Other: Placebo IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod
Other: Placebo IV — Intravenous infusion of placebo
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to measure the efficacy and safety of efgartigimod IV compared to placebo in participants with Acetylcholine Receptor Binding Antibody (AChR-Ab) seronegative Generalized Myasthenia Gravis (gMG). The study consists of a Part A where participants will be randomized to receive either efgartigimod IV or placebo IV and a Part B where participants completing part A will receive open-label efgartigimod IV. Participants will be in the study for up to (approximately) 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* The participant is at least 18 years of age and the local legal age of consent for clinical studies when signing the ICF.
* The participant is capable of providing signed informed consent and following with protocol requirements.
* The participant agrees to use contraceptive measures consistent with local regulations and the women of child-bearing potential (WOCBP) must have a negative serum pregnancy test result at screening and a negative urine pregnancy test result at baseline before receiving the study drug.
* The participant has no known weakness in infancy and later develop fatigable weakness after aged 16 years and diagnosed with acquired gMG of both of the following:

  1. History of abnormal neuromuscular transmission demonstrated by single fiber electromyography or repetitive nerve stimulation (RNS) or is anti-muscle-specific kinase antibodies (MuSK-Ab) seropositive
  2. Either a history of positive edrophonium chloride test OR a demonstrated improvement in MG signs with treatments such as oral acetylcholinesterase (AChE) inhibitors, plasma exchange (PLEX), immunoabsorption, or intravenous immunoglobulin (IVIg)/ subcutaneous immunoglobulin (SCIg) treatment
* The participant is receiving a stable dose of MG therapy before screening that includes acetylcholinesterase (AChE) inhibitors, steroids, or nonsteroidal immunosuppressive therapies (NSISTs) in combination or alone.

Exclusion Criteria:

* Known autoimmune disease or any medical condition that would interfere with an accurate assessment of clinical symptoms of gMG or puts the participant at undue risk
* History of malignancy, cancer, unless considered cured by adequate treatment with no evidence of recurrence for ≥3 years. Adequately treated participants with the following cancers can be included at any time: Basal cell or squamous cell skin cancer, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histological findings of prostate cancer
* Clinically significant active infection that is not sufficiently resolved in the investigator's opinion or positive serum test at screening for active infection with any of the following: Hepatitis B virus (HBV), Hepatitis C virus (HCV), HIV
* History of or current alcohol, drug, or medication abuse as assessed by the investigator
* Pregnant or lactating state or intention to become pregnant during the study
* Live or live-attenuated vaccine received <4 weeks before screening
* Worsening muscle weakness secondary to concurrent infections or medications
* Received a thymectomy less than 3 months before screening or thymectomy is planned during the study

The complete list of exclusion criteria can be found in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
MG-ADL total score change from baseline | Up to 29 days (part A)
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms)

SECONDARY OUTCOMES:
QMG total score change from baseline | Up to 8 weeks (part A) + 2 years (part B)
  The Quantitative myasthenia gravis (QMG) includes 13 items that measure endurance or fatigability and accounts for fluctuations in disease state. The total score ranges from 0 (no disease severity) to 39 (highest disease severity)
Proportion of participants who are both MG-ADL and QMG responders in part A | Up to 8 weeks (part A)
Proportion of participants with MSE | Up to 8 weeks (part A) + 2 years (part B)
  Minimal symptom expression (MSE) is defined as an MG-ADL total score of 0 or 1
Proportion of participants who are MG-ADL responders in part A | Up to 8 weeks (part A)
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms).
Proportion of participants who are QMG responders in part A | Up to 8 weeks (part A)
  The Quantitative myasthenia gravis (QMG) includes 13 items that measure endurance or fatigability and accounts for fluctuations in disease state. The total score ranges from 0 (no disease severity) to 39 (highest disease severity)
Proportion of participants who are early MG-ADL responders in part A | Up to 8 weeks (part A)
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms).
MG-ADL total score change from baseline over time in part A and part A+B | Up to 8 weeks (part A) + 2 years (part B)
  The Myasthenia Gravis Activities of Daily Living (MG- ADL) scale is an 8-item instrument used to assess MG symptoms and their effects on daily activities. The total score ranges from 0 (normal symptoms) to 24 (most severe symptoms).
MG-QoL15r change from baseline over time in part A and part A+B | Up to 8 weeks (part A) + 2 years (part B)
  The Myasthenia Gravis Quality of Life-15 revised (MG-QoL15r) is a patient-reported instrument that measures the impact of MG symptoms on quality of life. The total scores range from 0 (best outcome) to 30 (worst outcome)
EQ-5D-5L VAS change from baseline over time in part A and part A+B | Up to 8 weeks (part A) + 2 years (part B)
  The EQ-5D-5L is a participant-reported measure of health status developed by the EuroQol Group. The questionnaire comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Current health status is rated on vertical visual analog score (VAS) from 0 to 100, with a score of 0 corresponding to "the worst health you can imagine" and 100 corresponding to "the best health you can imagine."
Incidence of AEs and SAEs in part A and part A+B | Up to 8 weeks (part A) + 2 years (part B)
  AE: adverse event; SAE: serious adverse event
Total IgG concentrations percent changes from baseline over time in part A and part A+B | Up to 8 weeks (part A) + 2 years (part B)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (19):
  - HonorHealth Neurology - Bob Bove Neuroscience Institute, Scottsdale, Arizona
  - Loma Linda University Health, Fresno, California
  - First Choice Neurology Boca Raton, Boca Raton, Florida
  - SFM Clinical Research LLC, Boca Raton, Florida
  - The Neurology Institute / Healthcare Innovations Institute - Coral Springs, Coral Springs, Florida
  - Neurology Associates PA, Maitland, Florida
  - Desai Sethi Medical Center, Miami, Florida
  - Medsol Clinical Research Center Inc, Port Charlotte, Florida
  - BayCare - St. Anthony's Hospital, St. Petersburg, Florida
  - University of South Florida (USF) Health - Morsani Center for Advanced Healthcare, Tampa, Florida
  - Wellstar - Augusta University Medical Center, Augusta, Georgia
  - Kansas University Medical Center - Kansas City, Fairway, Kansas
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke University School of Medicine - Duke Early Phase Clinical Research Unit, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Erlanger Neuroscience Institute, Chattanooga, Tennessee
  - National Neuromuscular Research Institute, Austin, Texas
  - University of Washington Medical Center - Montlake, Seattle, Washington
- Belgium (4):
  - Hôpital Erasme, Anderlecht
  - Cliniques Universitaires Saint-Luc, Brussels
  - AZ Sint-Lucas Gent, Ghent
  - UZ Leuven, Leuven
- Canada (3):
  - Heritage Medical Research Clinic, Calgary
  - Genge Partners Inc., Montreal
  - Ottawa Hospital - Civic Campus, Ottawa
- China (14):
  - Xuanwu Hospital Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital of Guangxi Medical University, Guangxi
  - The First Affiliated Hospital of Guangzhou University Chinese Medicine, Guangzhou
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Qilu Hospital of Shandong University, Qingdao
  - Huashan Hospital Fudan University, Shanghai
  - First Hospital of Shanxi Medical University, Taiyuan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- Cyprus Institute of Neurology and Genetics, Égkomi, Cyprus
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Nemocnice Pardubickeho kraje, a.s., Pardubicka nemocnice, Pardubice
- Denmark (3):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense C
- Turun Yliopistollinen Keskussairaala, Turku, Finland
- France (3):
  - AP-HM- Hôpital de La Timone, Marseille
  - CHU de Nice-Hôpital Pasteur, Nice
  - AP-HP - Hôpital de la Pitié Salpétrière, Paris
- Georgia (5):
  - West Georgia Medical Center, Kutaisi
  - Petre Sarajishvili Institute of Neurology, Tbilisi
  - Pineo Medical Ecosystem, Tbilisi
  - New Hospitals, Tbilisi
  - LLC Caucasus Medical Centre, Tbilisi
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Katholisches Klinikum Bochum - St. Josef Hospital, Bochum
  - Universitätsklinikum Würzburg, Würzburg
- Greece (4):
  - Eginitio Hospital, Athens
  - University General Hospital ''ATTIKON'', Chaïdári
  - University General Hospital of Patras, Pátrai
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
- Semmelweis Egyetem Genomikai Medicina és Ritka Betegségek Intézete, Budapest, Hungary
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum Utrecht, Utrecht
- Norway (2):
  - Haukeland Universitetssykehus, Bergen
  - Oslo Universitetssykehus HF, Ullevål, Oslo
- Poland (6):
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Centrum Medyczne Neurologia Slaska, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
  - Krakowska Akademia Neurologii Sp. z o.o., Krakow
  - CLINIREM Sp z o.o., Lublin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu, Wroclaw
- Portugal (3):
  - ULS de Santa Maria, EPE - Hospital de Santa Maria, Lisbon
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Hospital de Santo António - Unidade Local de Saúde de Santo António, Porto
- Romania (2):
  - Cluj County Emergency Clinical Hospital, Cluj-Napoca
  - Sibiu Emergency County Clinical Hospital, Sibiu
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - National Guard Riyadh, Riyadh
- Serbia (2):
  - Opsta bolnica MSB - Medicinski Sistemi Beograd, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
- Spain (7):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (2):
  - Panthera Biopartners, Glasgow
  - Leeds General Infirmary, Leeds

REFERENCES:
- See also: US patient website — https://adaptseron.com/
- See also: US HCP website — https://adaptseronhcp.com/